CLINICAL TRIAL: NCT01412879
Title: A Randomized Phase II Trial of R-HCVAD/MTX/ARA-C Induction Followed by Consolidation With an Autologous Stem Cell Transplant Vs. R-Bendamustine Induction Followed by Consolidation With an Autologous Stem Cell Transplant for Patients ≤ 65 Years of Age With Previously Untreated Mantle Cell Lymphoma
Brief Title: S1106 Rituximab With Combination Chemotherapy or Bendamustine Hydrochloride Followed by Consolidation Chemotherapy and Stem Cell Transplantation in Older Patients With Previously Untreated Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000707601; S1106 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2011-08-06; First posted 2011-08-09 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Lymphoma
Keywords: contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Rituximab; Bendamustine Hydrochloride; Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Leucovorin; Methotrexate; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Course 1 and 3: Patients receive induction therapy comprising rituximab IV on day 1; cyclophosphamide IV over 3 hours every 12 hours on days 2-4; doxorubicin hydrochloride IV over 72 hours on days 5-7; vincristine sulfate IV on days 5 and 12; and dexamethasone IV or orally (PO) once daily (QD) on days 2-5 and 12-15. Patients with responsive disease after course 1 proceed to course 2. Course 2 and 4: Patients receive rituximab IV on day 1; methotrexate IV over 2-22 hours on day 2; cytarabine IV over 2 hours every 12 hours on days 3-4; and leucovorin calcium PO or IV on days 3-6. Patients then undergo stem cell collection after completion of course 2. Patients undergo stem cell collection after completion of course 2.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: leucovorin calcium; Drug: methotrexate; Drug: vincristine sulfate
- Arm II (Experimental): Course 1-6: Patients receive rituximab IV on day 1 and bendamustine hydrochloride IV over 30 minutes on days 1-2. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Beginning 3-4 weeks later, patients with responsive disease receive 2 additional courses of treatment. Beginning within 8 weeks, patients receive rituximab IV and cyclophosphamide IV over 1 hour on day 1. Patients then undergo stem cell collection about 26 days later.
  Interventions: Biological: rituximab; Drug: bendamustine hydrochloride; Drug: cyclophosphamide

INTERVENTIONS:
Biological: rituximab — Given IV
Drug: bendamustine hydrochloride — Given IV
  Arms: Arm II
Drug: cyclophosphamide — Given IV
Drug: cytarabine — Given IV
  Arms: Arm I
Drug: dexamethasone — Given PO or IV
  Arms: Arm I
Drug: doxorubicin hydrochloride — Given IV
  Arms: Arm I
Drug: leucovorin calcium — Given PO or IV
  Arms: Arm I
Drug: methotrexate — Given IV
  Arms: Arm I
Drug: vincristine sulfate — Given IV
  Arms: Arm I

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and help kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy also work in different ways to kill more cancer cells or stop them from growing. It is not yet known whether rituximab is more effective with combination chemotherapy or bendamustine hydrochloride in treating patients with mantle cell lymphoma undergoing peripheral blood stem cell transplantation.

PURPOSE: This randomized phase II trial studies how well giving rituximab together with combination chemotherapy or bendamustine hydrochloride followed by consolidation chemotherapy and peripheral blood stem cell transplantation works in treating older patients with previously untreated mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To estimate the 2-year progression-free survival (PFS) of patients with newly diagnosed mantle cell lymphoma (MCL) treated with rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, dexamethasone (RHCVAD), methotrexate and cytarabine (MTX/Ara-C), and autologous stem cell transplant (ASCT) or rituximab and bendamustine (R-bendamustine) and autologous stem cell transplant and to select a regimen for further development.
* To assess the response rate and overall survival of patients with newly diagnosed MCL treated with R-HCVAD/MTX/Ara-C and ASCT or R-bendamustine and ASCT.
* To assess the toxicity and tolerability of R-HCVAD/MTX/Ara-C and ASCT or R-bendamustine and ASCT in patients with newly diagnosed MCL.
* To determine the prognostic value of quantitative minimal-residual disease (MRD) monitoring in the peripheral blood of MCL patients after induction therapy and serially after high-dose chemotherapy and ASCT on treatment outcome.
* To bank diagnostic tissue sections for future translational research studies.

OUTLINE: This is a multicenter study. Patients are stratified according to risk classification by Mantle Cell Lymphoma International prognostic Index (MIPI) score (low risk vs intermediate/high risk). Patients are randomized to 1 of 2 treatment arms.

* Arm I (induction therapy):

  * Courses 1 and 3: Patients receive induction therapy comprising rituximab IV on day 1; cyclophosphamide IV over 3 hours every 12 hours on days 2-4; doxorubicin hydrochloride IV over 72 hours on days 5-7; vincristine sulfate IV on days 5 and 12; and dexamethasone IV or orally (PO) once daily (QD) on days 2-5 and 12-15. Patients with responsive disease after course 1 proceed to course 2.
  * Course 2 and 4: Patients receive rituximab IV on day 1; methotrexate IV over 2-22 hours on day 2; cytarabine IV over 2 hours every 12 hours on days 3-4; and leucovorin calcium PO or IV on days 3-6. Patients undergo stem cell collection after completion of course 2.
  * Each course is 21 days long and continues in the absence of disease progression or unacceptable toxicity.
* Arm II (induction therapy):

  * Course 1-6: Patients receive rituximab IV on day 1 and bendamustine hydrochloride IV over 30 minutes on days 1-2. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Beginning 3-4 weeks later, patients with responsive disease receive 2 additional courses of treatment.
  * Stem cell mobilization: Beginning within 8 weeks, patients receive rituximab IV and cyclophosphamide IV over 1 hour on day 1. Patients then undergo stem cell collection about 26 days later.

Consolidation therapy: Patients receive one of the following preparative regimens.

* BCV* chemotherapy: Carmustine IV over 2 hours on days -6 to -4; etoposide IV over 4 hours on day -4; and cyclophosphamide IV over 1 hour on day -2.
* BEAM* chemotherapy: Carmustine IV over 4 hours on days -7 and -6; etoposide IV over 1 hour twice daily and cytarabine IV over 2 hours twice daily on days -5 to -2, and melphalan IV on day -1.
* TBI, etoposide, cyclophosphamide: Patients undergo total-body irradiation (TBI)** twice daily on days -8 to -5. Patients also receive etoposide IV on day -4 and cyclophosphamide IV over 1 hour on day -2.
* NOTE: * Patients 61 years of age or older receive either BCV or BEAM.
* NOTE: * *TBI may not be used for patients 61 years of age and older. Stem cell transplantation: Patients then undergo autologous peripheral blood stem cell transplantation on day 0.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 2 years, and then annually for up to 8 years from registration.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* All patients must have previously untreated stage III, IV, or bulky stage II mantle cell lymphoma (MCL)

  * A diagnosis of MCL must be confirmed by histopathological diagnosis including immunohistochemistry and flow cytometry documenting both of the following phenotypes:

    * CD19+ or CD20+
    * Cyclin D1+ or evidence of the t(11;14) translocation by cytogenetics or FISH
* Adequate sections from the original diagnostic specimen must be available for submission for central review

  * An adequate biopsy requires sufficient tissue to establish the architecture and a WHO histologic subtype with certainty

    * Core biopsies, especially multiple core biopsies, MAY be adequate, but needle aspirations or cytologies are not adequate
  * Bone marrow core biopsy or clot sections (not aspirates) may be used as diagnostic material if it is significantly involved and are the only diagnostic material available
* All patients must have bidimensional measurable disease documented on the Lymphoma Baseline Tumor Assessment Form (Form #48031)

  * Patients who also have non-measurable disease in addition to measurable disease must have all nonmeasurable disease assessed within 28 days prior to registration
* Patients must not have clinical evidence of central nervous system (CNS) involvement by lymphoma

  * Any laboratory or radiographic tests performed prior to registration to assess CNS involvement must be negative
* Patients must have a unilateral/bilateral bone marrow aspirate and biopsy for staging performed within 42 days prior to registration

  * If the biopsy cannot be performed but the aspirate is unequivocally consistent with mantle cell lymphoma, this will be considered adequate for staging purposes
* Patients must be eligible for stem cell transplantation by institutional guidelines with the plan that transplant will be conducted at a cooperative group-approved transplant center

  * Patients must be planning to undergo stem cell transplantation within 84 days after day 1 of the last induction course
  * Patients must have had at least 1.5 X 10^6 CD34^+ cells/kg collected and stored prior to second registration for stem cell transplantation

PATIENT CHARACTERISTICS:

* Zubrod performance status of 0-2
* Bilirubin ≤ 3 times upper limit of normal (ULN)
* Serum creatinine ≤ 2.0 times ULN
* Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Platelet count ≥ 100,000/mcL, unless due to bone marrow infiltration by lymphoma
* All patients ≥ 45 years of age must have an echocardiogram (ECHO) or Multi Gated Acquisition Scan (MUGA )scan within 42 days prior to registration (whichever method is used at baseline must be used at restaging)

  * Patients < 45 years of age should have ECHO/MUGA only if clinically indicated
  * Patients with an ejection fraction < institutional lower limit of normal (ILLN) are not eligible
* Serum Lactate dehydrogenase (LDH) and a Complete Blood Count (CBC with differential must be measured within 28 days prior to registration
* Patients known to be HIV positive, or who have a history of solid organ transplantation, are ineligible
* No active hepatitis
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer; in situ cervical cancer; adequately treated Stage I or II cancer from which the patient is currently in complete remission; or any other cancer from which the patient has been disease-free for 5 years
* Pregnant or nursing women may not participate
* Women or men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-11; Primary Completion 2016-02 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Bernstein, MD, Principal Investigator — James P. Wilmot Cancer Center
Locations (204):
- United States (204):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - St. Joseph Regional Medical Center, Lewiston, Idaho
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Union Hospital of Cecil County, Elkton, Maryland
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Baylor University Medical Center - Dallas, Dallas, Texas
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Swedish Medical Center - Issaquah Campus, Issaquah, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Northwest Cancer Specialists at Vancouver Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: R-HCVAD/MTX/Ara-C (Induction Therapy): The R-HCVAD/MTX/ARA-C combination are rituximab, cyclophosphamide, vincristine, doxorubicin, dexamethasone, methotrexate, and cytarabine. Cycle 1 and 3: Patients receive induction therapy comprising rituximab IV on day 1; cyclophosphamide IV over 3 hours every 12 hours on days 2-4; doxorubicin hydrochloride IV over 72 hours on days 5-7; vincristine sulfate IV on days 5 and 12; and dexamethasone IV or orally (PO) once daily (QD) on days 2-5 and 12-15. Patients with responsive disease after course 1 proceed to course 2. Cycle 2 and 4: Patients receive rituximab IV on day 1; methotrexate IV over 2-22 hours on day 2; cytarabine IV over 2 hours every 12 hours on days 3-4; and leucovorin calcium PO or IV on days 3-6. Patients undergo stem cell collection after completion of Cycle 2 (1 cycle = 21 days).
- Arm 2: R-Bendamustine (Induction Therapy): R-bendamustine combinations are rituximab and bendamustine. Patients receive rituximab IV on day 1 and bendamustine hydrochloride IV over 30 minutes on days 1-2. Treatment repeats every 28 days for 4 cycles (1 cycle = 28 days). Patients with responsive disease receive 2 additional cycles of treatment. Patients undergo stem cell collection after completion of 6 Cycles of treatment.
- Consolidation Therapy: Stem Cell Transplant: Patients receive stem cell transplant with non-TBI containing regimen (BCV or BEAM Chemotherapy) for patients 61 years or older or TBI-containing regimen (TBI/VP-16/Cyclophosphamide). BCV chemotherapy: Carmustine IV over 2 hours on days -6 to -4; etoposide IV over 4 hours on day -4; and cyclophosphamide IV over 1 hour on day -2. BEAM chemotherapy: Carmustine IV over 4 hours on days -7 and -6; etoposide IV over 1 hour twice daily and cytarabine IV over 2 hours twice daily on days -5 to -2, and melphalan IV on day -1.
  TBI, etoposide, cyclophosphamide: Patients undergo total-body irradiation (TBI)** twice daily on days -8 to -5. Patients also receive etoposide IV on day -4 and cyclophosphamide IV over 1 hour on day -2. * *TBI may not be used for patients 61 years of age and older. Stem cell transplantation: Patients then undergo autologous peripheral blood stem cell transplantation on day 0.
Period: Initial Registration (Induction Therapy)
Arm/Group | Arm 1: R-HCVAD/MTX/Ara-C (Induction Therapy) | Arm 2: R-Bendamustine (Induction Therapy) | Consolidation Therapy: Stem Cell Transplant
Started | 18 | 35 | 0
Treatment Started | 17 | 35 | 0
Completed | 5 | 27 | 0
Not Completed | 13 | 8 | 0
Not completed — Adverse Event | 5 | 3 | 0
Not completed — Refusal Unrelated to Adverse Event | 1 | 3 | 0
Not completed — Progression/Relapse | 0 | 1 | 0
Not completed — Reasons not Protocol Specified | 6 | 1 | 0
Not completed — Treatment not Given | 1 | 0 | 0
Period: Consolidation Therapy
Arm/Group | Arm 1: R-HCVAD/MTX/Ara-C (Induction Therapy) | Arm 2: R-Bendamustine (Induction Therapy) | Consolidation Therapy: Stem Cell Transplant
Started | 0 | 0 | 26 (Only eligible patients who are able to have stem cell harvested receive consolidation therapy.)
Completed | 0 | 0 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients who started treatment were included in the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: R-HCVAD/MTX/Ara-C (Induction Therapy) | Arm 2: R-Bendamustine (Induction Therapy) | Total
Number analyzed (Participants) | 17 | 35 | 52
Age, Continuous [Median (Full Range); unit: years] | 58.8 [43.6 to 65.7] | 56.6 [33.0 to 64.1] | 57.2 [33.0 to 65.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 9 | 32 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 35 | 51
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 13 | 32 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) at 2 Years
Description: Disease progression is defined using the 2007 revised Cheson et al. criteria that is at least 50% increase in sum of the product of the diameters (SPD) of target measurable nodal lesions over the smallest sum observed, or >= 50% increase in greatest transverse diameter (GTD) of any nodal > 1 cm in shortest axis, or >= 50% increase in the SPD of other target measurable lesions over the smallest sum observed, any new bone marrow involvement, any new lesion, lymph node with long axis is > 1.5 cm or if both long and short axes are > 1 cm, PET positive if patients with no pretreatment PET scan or when PET scan was positive before therapy. Progression-free survival is measured from date of registration to date of first observation of progressive disease, or death due to any cause. Patients last known to be alive and progression-free are censored at date of last contact.
Time Frame: Up to 2 years
Population: All eligible patients who started treatment were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: R-HCVAD/MTX/Ara-C (Induction Therapy) | Arm 2: R-Bendamustine (Induction Therapy)
Number analyzed (Participants) | 17 | 35
percentage of participants | 82 [53.0 to 93.7] | 81 [62.7 to 91.1]

2. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Up to 8 months (Assessed at the beginning of each cycle of treatment, at restaging, and at post transplant.)
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 4.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Groups:
- R-HCVAD/MTX/Ara-C (Induction Therapy): The R-HCVAD/MTX/ARA-C combination are rituximab, cyclophosphamide, vincristine, doxorubicin, dexamethasone, methotrexate, and cytarabine. Cycle 1 and 3: Patients receive induction therapy comprising rituximab IV on day 1; cyclophosphamide IV over 3 hours every 12 hours on days 2-4; doxorubicin hydrochloride IV over 72 hours on days 5-7; vincristine sulfate IV on days 5 and 12; and dexamethasone IV or orally (PO) once daily (QD) on days 2-5 and 12-15. Patients with responsive disease after course 1 proceed to course 2. Cycle 2 and 4: Patients receive rituximab IV on day 1; methotrexate IV over 2-22 hours on day 2; cytarabine IV over 2 hours every 12 hours on days 3-4; and leucovorin calcium PO or IV on days 3-6. Patients undergo stem cell collection after completion of Cycle 2 (1 cycle = 21 days).
- R-Bendamustine (Induction Therapy): R-bendamustine combinations are rituximab and bendamustine. Patients receive rituximab IV on day 1 and bendamustine hydrochloride IV over 30 minutes on days 1-2. Treatment repeats every 28 days for 4 cycles (1 cycle = 28 days). Patients with responsive disease receive 2 additional cycles of treatment. Patients undergo stem cell collection after completion of 6 Cycles of treatment.
- Stem Cell Transplant (Consolidation Therapy): Patients receive stem cell transplant with non-TBI containing regimen (BCV or BEAM Chemotherapy) for patients 61 years or older or TBI-containing regimen (TBI/VP-16/Cyclophosphamide). BCV chemotherapy: Carmustine IV over 2 hours on days -6 to -4; etoposide IV over 4 hours on day -4; and cyclophosphamide IV over 1 hour on day -2. BEAM chemotherapy: Carmustine IV over 4 hours on days -7 and -6; etoposide IV over 1 hour twice daily and cytarabine IV over 2 hours twice daily on days -5 to -2, and melphalan IV on day -1.
  TBI, etoposide, cyclophosphamide: Patients undergo total-body irradiation (TBI)** twice daily on days -8 to -5. Patients also receive etoposide IV on day -4 and cyclophosphamide IV over 1 hour on day -2. * *TBI may not be used for patients 61 years of age and older. Stem cell transplantation: Patients then undergo autologous peripheral blood stem cell transplantation on day 0.
Arm/Group | R-HCVAD/MTX/Ara-C (Induction Therapy) | R-Bendamustine (Induction Therapy) | Stem Cell Transplant (Consolidation Therapy)
Number analyzed (Participants) | 17 | 35 | 26
Participants
  Acidosis | 0 | 0 | 1
  Adult respiratory distress syndrome | 0 | 0 | 1
  Alanine aminotransferase increased | 1 | 0 | 0
  Anemia | 10 | 3 | 9
  Anorexia | 0 | 0 | 1
  Arthralgia | 0 | 1 | 0
  Aspartate aminotransferase increased | 1 | 0 | 0
  Blood bilirubin increased | 0 | 0 | 2
  CD4 lymphocytes decreased | 2 | 2 | 0
  Catheter related infection | 1 | 1 | 1
  Dehydration | 1 | 0 | 0
  Device related infection | 0 | 0 | 1
  Diarrhea | 1 | 0 | 4
  Enterocolitis | 0 | 0 | 1
  Enterocolitis infectious | 0 | 1 | 1
  Epistaxis | 1 | 0 | 0
  Fatigue | 0 | 1 | 0
  Febrile neutropenia | 5 | 5 | 13
  Gallbladder infection | 0 | 0 | 1
  Hyperglycemia | 2 | 0 | 0
  Hypoalbuminemia | 0 | 1 | 0
  Hypocalcemia | 0 | 0 | 2
  Hypokalemia | 5 | 2 | 1
  Hypomagnesemia | 0 | 0 | 1
  Hyponatremia | 0 | 0 | 1
  Hypophosphatemia | 4 | 1 | 3
  Hypotension | 0 | 0 | 1
  Hypoxia | 0 | 0 | 1
  Infections and infestations - Other, specify | 0 | 1 | 0
  Infusion related reaction | 0 | 1 | 0
  Lung infection | 0 | 0 | 1
  Lymphocyte count decreased | 10 | 27 | 12
  Myalgia | 0 | 1 | 0
  Nausea | 1 | 0 | 2
  Neutrophil count decreased | 11 | 12 | 16
  Pain in extremity | 0 | 1 | 0
  Platelet count decreased | 12 | 6 | 19
  Pruritus | 0 | 1 | 0
  Rash maculo-papular | 1 | 1 | 1
  Rectal hemorrhage | 0 | 0 | 1
  Small intestinal obstruction | 0 | 0 | 1
  Sore throat | 0 | 1 | 0
  Syncope | 1 | 0 | 0
  Tumor pain | 0 | 1 | 0
  Urinary tract infection | 0 | 1 | 0
  Vascular access complication | 0 | 1 | 0
  Vomiting | 0 | 0 | 1
  White blood cell decreased | 10 | 14 | 20

3. Secondary Outcome: Response Rate (Complete and Partial Response)
Description: Complete Response (CR) is a complete disappearance of all disease with the exception of the following. If no PET scan or when the PET scan was positive before therapy, a post-treatment residual mass of any size is permitted if it is PET negative. If the PET scan was negative before therapy, all nodal masses at baseline must have regressed. No new lesions. Previously enlarged organs must have regressed and not be palpable. Bone marrow (BM) must be negative if positive at baseline. Normalization of markers. Partial Response (PR) is a 50% decrease in the sum of products of greatest diameters (SPD) for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes. If PET scan or when the PET scan was positive before therapy, PET should be positive in at least one previously involved site.
Time Frame: Up to 9 months
Population: All eligible patients who started treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: R-HCVAD/MTX/Ara-C (Induction Therapy) | Arm 2: R-Bendamustine (Induction Therapy)
Number analyzed (Participants) | 17 | 35
percentage of participants | 94.1 [71.3 to 99.9] | 82.9 [66.4 to 93.4]

4. Secondary Outcome: 5-year Overall Survival (OS)
Description: Measured from date of registration to date of death due to any cause. Patients last known to be alive and are censored at date of last contact.
Time Frame: Up to 5 years
Population: All eligible patients who started treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: R-HCVAD/MTX/Ara-C (Induction Therapy) | Arm 2: R-Bendamustine (Induction Therapy)
Number analyzed (Participants) | 17 | 35
percentage of participants | 81 [50.6 to 93.3] | 79 [57.1 to 90.1]

ADVERSE EVENTS:
Time Frame: Up to 8 months (assessed at the beginning of each cycle of treatment, at restaging, and at post transplant).
Arm/Group | R-HCVAD/MTX/Ara-C (Induction Therapy) | R-Bendamustine (Induction Therapy) | Stem Cell Transplant (Consolidation Therapy)
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/35 | 1/26
Other Adverse Events (participants affected / at risk) | 17/17 | 35/35 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R-HCVAD/MTX/Ara-C (Induction Therapy) (N=17) | R-Bendamustine (Induction Therapy) (N=35) | Stem Cell Transplant (Consolidation Therapy) (N=26)
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R-HCVAD/MTX/Ara-C (Induction Therapy) (N=17) | R-Bendamustine (Induction Therapy) (N=35) | Stem Cell Transplant (Consolidation Therapy) (N=26)
Anemia (Blood and lymphatic system disorders) | 15 | 25 | 21
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 5 | 13
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 3 | 1
Sinus tachycardia (Cardiac disorders) | 3 | 3 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Blurred vision (Eye disorders) | 0 | 3 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Watering eyes (Eye disorders) | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 3
Anal pain (Gastrointestinal disorders) | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 12 | 16 | 4
Diarrhea (Gastrointestinal disorders) | 8 | 10 | 20
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 2
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 2
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 2 | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 7 | 2 | 13
Nausea (Gastrointestinal disorders) | 9 | 22 | 19
Rectal pain (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 4 | 8 | 9
Chills (General disorders) | 2 | 4 | 1
Edema face (General disorders) | 1 | 0 | 0
Edema limbs (General disorders) | 2 | 4 | 5
Facial pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 11 | 33 | 15
Fever (General disorders) | 0 | 9 | 4
Infusion related reaction (General disorders) | 3 | 4 | 0
Irritability (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 2 | 0
Pain (General disorders) | 1 | 6 | 0
Allergic reaction (Immune system disorders) | 0 | 3 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 1 | 1
Infections and infestations-Other (Infections and infestations) | 1 | 5 | 0
Lung infection (Infections and infestations) | 0 | 0 | 2
Skin infection (Infections and infestations) | 0 | 2 | 2
Upper respiratory infection (Infections and infestations) | 0 | 3 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 2 | 0
Alanine aminotransferase increased (Investigations) | 8 | 8 | 7
Alkaline phosphatase increased (Investigations) | 3 | 7 | 4
Aspartate aminotransferase increased (Investigations) | 4 | 9 | 6
Blood bilirubin increased (Investigations) | 1 | 7 | 5
CD4 lymphocytes decreased (Investigations) | 2 | 2 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 1 | 0 | 0
Cholesterol high (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 3 | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 1 | 0
INR increased (Investigations) | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 11 | 29 | 14
Neutrophil count decreased (Investigations) | 11 | 18 | 18
Platelet count decreased (Investigations) | 15 | 23 | 19
Weight gain (Investigations) | 1 | 3 | 2
Weight loss (Investigations) | 1 | 4 | 3
White blood cell decreased (Investigations) | 11 | 24 | 20
Anorexia (Metabolism and nutrition disorders) | 6 | 12 | 12
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 14 | 8
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 4 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 4 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 7 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 8 | 17
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 7 | 7 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 2 | 5
Hyponatremia (Metabolism and nutrition disorders) | 5 | 8 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 3 | 4
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 7 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 7 | 2
Cognitive disturbance (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 5 | 0
Dysgeusia (Nervous system disorders) | 2 | 3 | 4
Headache (Nervous system disorders) | 6 | 6 | 3
Nervous system disorders-Other (Nervous system disorders) | 0 | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 2 | 3
Presyncope (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 3 | 6 | 1
Depression (Psychiatric disorders) | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 6 | 3
Proteinuria (Renal and urinary disorders) | 1 | 1 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 3 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 11 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 3 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 9 | 2
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 4 | 1
Flushing (Vascular disorders) | 1 | 0 | 1
Hot flashes (Vascular disorders) | 0 | 3 | 0
Hypertension (Vascular disorders) | 2 | 11 | 5
Hypotension (Vascular disorders) | 2 | 6 | 6
Thromboembolic event (Vascular disorders) | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No